CLINICAL TRIAL: NCT03477669
Title: Infantile Colic: A Prospective, Randomized, Double Blind, Placebo Controlled Study of the Efficacy of Lactobacillus GG (ATCC 53103) Plus Chamomile in Breastfeeding Infants
Brief Title: Infantile Colic: Study of the Efficacy of Lactobacillus GG (ATCC 53103) Plus Chamomile in Breastfeeding Infants
Acronym: Colic
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit study participants
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0060-18-FB
Record Dates: First submitted 2018-03-07; First posted 2018-03-26 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Infantile Colic
Keywords: Colic
MeSH Terms: conditions — Colic | interventions — Chamomile extract

STUDY DESIGN:
Intervention Model Description: The study will be performed as a 4 week, placebo controlled, pilot trial with a one week run in period. Thirty subjects will be randomly assigned to each group for a total enrollment of 60 infants.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chamomile/probiotic arm (Experimental): Infant will receive 5 drops of the study product once per day with a feeding at midday.
  Interventions: Dietary Supplement: chamomile/probiotic arm
- Placebo of chamomile/probiotic arm (Placebo Comparator): Infant will receive 5 drops of a placebo product once a day at midday.
  Interventions: Dietary Supplement: Placebo of chamomile/probiotic arm

INTERVENTIONS:
Dietary Supplement: chamomile/probiotic arm — Caregivers will administer 5 drops of the study product once a day with a feeding at mid-day.
  Arms: chamomile/probiotic arm
Dietary Supplement: Placebo of chamomile/probiotic arm — Caregivers will administer 5 drops of the placebo study product once a day with a feeding at mid-day.
  Arms: Placebo of chamomile/probiotic arm

SUMMARY:
The objective of this study is to determine the efficacy of a product combining the probiotic Lactobacillus GG and chamomile in treating infantile colic in exclusively breast fed infants. The study will be performed as a 4 week, placebo controlled, pilot trial with a one week run in period. Thirty subjects will be randomly assigned to each group for a total enrollment of 60 infants.

DETAILED DESCRIPTION:
The study will be performed as a 4 week, placebo controlled, pilot trial with a one week run in period. Thirty participants will be randomly assigned to each group for a total enrollment of 60 participants. Participants will be recruited from the Children's' Hospital & Medical Center's Pediatrician's group. The study coordinators and Investigators will conduct informational lunches at selected pediatrician offices in the Omaha area. The investigators will introduce the topic of the colic study to participants seen for routine follow up who the investigators suspect may meet the diagnostic criteria for colic. The study coordinator will then contact the participants and assess suitability with a brief phone questionnaire. If participants appear to qualify and the participant is agreeable an enrollment appointment will be made to sign the consent, education on the product and how to administer it, teaching regarding diary instrument and completion of the quality of life survey. A brief medical history including the delivery mode and family allergy history will be collected as well as weight and length of the infant at the consent visit. A subset of participants will be asked to provide a stool sample for analysis of calprotectin level (a marker of intestinal inflammation) if the participants are willing to provide this. Participants will administer 5 drops of the study product once a day with a feeding at mid-day. Participants will be instructed to record crying time for a 1 week run in period and then administer the provided drops as directed once a day and record daily crying time on 3 days each week for 4 subsequent weeks. A follow up phone call 2 weeks after starting the product will be conducted to ensure compliance and assess for any adverse events. A final visit after 4 weeks will be conducted for collection of the diary data, completion of the quality of life survey, obtainment of the infant's length and weight and collection of a follow up stool sample if the provided one at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver is able to give written informed assent and willingness to participate in the study and comply with its procedures
* Male or Female
* Born at term (38-41 weeks gestation)
* Aged 3 wks-16 wks
* Be in generally good health as determined by the investigators
* BMI between 5th and 95th percentiles
* Exclusively breastfeeding throughout the study
* Be willing to complete crying diary
* Be willing to administer the probiotic as prescribed
* Be willing to completed the Quality of Life instrument before and after the intervention
* Meets the Rome criteria for colic

Exclusion Criteria:

* Are less than 3 weeks or greater than 17 weeks of age or older
* Underweighted or obese based on BMI. Less than 5th or greater than 95th percentiles
* Mothers on an exclusively vegan diet and those with a chronic disease requiring medication therapy
* Mothers or infants having a significant acute or chronic existing illness [cardiovascular, gastrointestinal, immunological] or a condition, which in the investigators judgment contraindicates involvement in the study
* Mothers or infants having a condition or taking a medication, dietary supplement or food product that the investigator believes would interfere with the objectives of the study pose a safety risk or confound the interpretation of the study results
* Individuals who, in the opinion of the investigator, are considered to be poor clinical attendees or unlikely for any reason to be able to comply with the trial
* Mothers or infants who are receiving treatment involving experimental drugs
* Participation in a recent experimental trial less than 30 days prior to this study
* Inability to complete the diary, survey scales and appointments
* First degree relative allergic to ragweed, asters, or chrysanthemums
* The following concomitant medications are not allowed at any time during or 1 week prior to initiation of the study: antibiotics or probiotics

Ages: 3 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Crying time | 4 weeks
  The investigators will be comparing time on the Baby's Day Diary © from the 1 week run-in to the end of the 4 week period and hope to see a 50% drop in crying time listed on the Baby's Day Diary© .

SECONDARY OUTCOMES:
Quality of Life-The Short Form -36 (SF-36) | 4 weeks
  Measurement of QOL scores before and after treatment with the drops. The investigators hope to see an improvement in the participants Qualify of Life scores over the 4 week study.
Calprotectin levels | 4 weeks
  The investigators hope to see a significant decrease in the baby's calprotectin stool levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ruben E Quiros, MD, Principal Investigator — University of Nebraska
Locations (1):
- Children's Hospital & Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No